CLINICAL TRIAL: NCT06905444
Title: Effects of Multimodal Therapy Versus Myofascial Release Techniques in Patient With Upper Cross Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/785
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Upper Extremity Dysfunction
MeSH Terms: interventions — Myofascial Release Therapy; Combined Modality Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial Release Technique (Experimental)
  Interventions: Combination Product: Myofascial Release Technique
- Multimodal Therapy (Active Comparator)
  Interventions: Combination Product: Multimodal Therapy

INTERVENTIONS:
Combination Product: Myofascial Release Technique — "GROUP A (Multimodal Therapy) Group A was treated with multimodal therapy for 30-45 minutes for 2 sessions per week for 6 weeks. Postural education like correct posture and forward head posture exercises like chin tuck in. Patient was sitting on chair. Therapist was standing on side of patient treated part. Strengthening exercises for the deep cervical flexors, shoulder blade stabilizers, and core muscles with 3 Sets of 3 repetitions with hold for 5 seconds of each exercise. Then breathing exercises for 1 minute. Then grade A (pain free range) cervical spine mobilization 1 Set of 3 repetition. During entire treatment session, the therapist kept close eye on patient's discomfort.
  Arms: Myofascial Release Technique
Combination Product: Multimodal Therapy — Group B (Myofascial Release Technique) Group B was treated with multimodal therapy for 30-45 minutes for 2 sessions per week for 6 weeks. Palpate the muscles and fascia to identify areas of restriction. Apply gentle, sustained pressure to the restricted area using the fingertips or knuckles for Fascial Unwinding. Hold the pressure for 3-5 minutes to allow the fascia to release. Encourage the patient to breathe deeply and slowly to promote relaxation. The stretching of tight muscles 1 set of 3 repetitions. Apply gentle, sustained pressure to release tension of these tight muscles, Suboccipital, Scalene, Pectoralis Major, Trapezius, Levator Scapulae
  Arms: Multimodal Therapy

SUMMARY:
Upper Cross Syndrome (UCS) is a frequent condition which is most commonly encountered in the musculoskeletal disorders showing a characteristics pattern of muscular imbalance and dysfunction in the joints of the neck and shoulder region. Upper Cross Syndrome remains a prevalent and debilitating condition, despite optimal approaches aimed at reducing pain and improving function.

DETAILED DESCRIPTION:
This study investigates the additional benefits of Multimodal Therapy and Myofascial Release Technique in individuals with Upper Cross Syndrome. Rooted .The researcher employs a randomized controlled trial methodology. Participants are divided into two groups: one receiving Multimodal Therapy, and the other receiving Myofascial Release Techniques. Outcomes are assessed over a 6-week period, focusing on pain levels, Posture and functional disability by goniometer, Numeric pain rating scale (NPRS), Neck disability index (NDI) scores and REEDCO posture assessment scale.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed by physician with sign and symptoms includes muscle in neck, chest and shoulder become overactive or underactive creating the X shape.
* Office worker.
* Aged 20 to 40 years.
* Male and females.

Exclusion Criteria:

* Recent trauma or surgery to the neck or shoulder region.
* Cancer or Metastasis in the neck or shoulder region.
* Infection or Abscess in the neck or shoulder region.
* Neurological conditions.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
NUMERIC PAIN RATING SCALE (NPRS) | 12 Months
  The 11-point numeric scale ranges from '0' representing "no pain" to feed '10' representing "pain as bad as you can imagine" or "worst pain imaginable".
NECK DIABILITY INDEX (NDI) | 12 Months
  The questionnaire has been designed to evaluate how cervical pain affects ability in managing daily routine functions. There are 10 sections includes 10 questions related to pain intensity, personal care, weight lifting, reading, headaches, concentration, work , driving, sleeping and recreations. Scale between 0-5 score. Total score is 50. 22% or more score is considering significant activities of daily living disability.
REEDCO POSTURE ASSESSMENT SCALE | 12 Months
  Standard tool for objective and quality measurement of postural deviation association with pictures. This includes name, sex, age, center, date and physiotherapist. The total score is out of 100. Normal range between 80-100% of ROM. Mild restriction 60-79% ROM.Moderate restriction 40-59% and Severe restriction: 0-39% ROM. Interpretation of scale is Good -10, Fair -5, Poor - 0 the assessment of muscle.

CONTACTS AND LOCATIONS:
Locations (1):
- Alkhidmat hospital Sahiwal, Sahiwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No